CLINICAL TRIAL: NCT06581588
Title: Apnoeic Oxygenation in Obstructive Sleep Apnea: a Randomised Controlled Trial Comparing Transnasal Humidified Rapid Insufflation Ventilator Exchange (THRIVE) Combined With Nasopharyngeal Airway and THRIVE Alone
Brief Title: Apneic Oxygenation by Transnasal Humidified Rapid Insufflation Ventilator Exchange Obstructive Sleep Apnea Patients
Acronym: THRIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TREC2024-KY069
Record Dates: First submitted 2023-08-18; First posted 2024-09-03 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2024-08

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: Obstructive sleep apnea; THRIVE; apnea time; nasopharyngeal; nasopharyngeal airway
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oxygenation using THRIVE technique (Active Comparator): oxygenation delivered via nasal high flow humidified oxygen (Optiflow) . 70 litres/minute
  Interventions: Device: THRIVE
- THRIVE combined nasopharyngeal airway (Experimental): oxygenation delivered via nasopharyngeal airway and THRIVE technique. 70 litres/minute
  Interventions: Device: THRIVE combine nasopharyngeal airway

INTERVENTIONS:
Device: THRIVE — Device: Optiflow and THRIVE technique Nasal high flow humidified oxygen
  Arms: oxygenation using THRIVE technique
Device: THRIVE combine nasopharyngeal airway — Device: Optiflow and THRIVE technique Nasal high flow humidified oxygen and nasopharyngeal airway
  Arms: THRIVE combined nasopharyngeal airway

SUMMARY:
The purpose of the study is to compare effectiveness of different methods of achieving oxygenation in obstructive sleep apnea patients. The investigators intend to compare transnasal humidified rapid-insufflation ventilator exchange (THRIVE) combined with nasopharyngeal airway with THRIVE alone.

DETAILED DESCRIPTION:
With the increasing prevalence of obesity, the prevalence of OSA is also rising, ranging from 9% to 25% in the general adult population. Patients with OSA have features of an anatomically tricky airway due to a crowded collapsible pharyngeal space, compounded by physiological problems related to lower functional residual capacity and increased oxygen consumption, leading to faster oxygen desaturation. Meanwhile, patients with OSA, compared to patients without OSA, have a 3-4 times higher risk of difficult intubation, difficult mask ventilation, or both. Apnoea time is a potentially hazardous period during induction of anesthesia and it is particularly so in patients with OSA. OSA patients undergoing general anesthesia gave rise to many concerns and challenges, and strategies to extend the apneic time were required. Identifying the most effective method of oxygenating OSA patients can therefore significantly improve the safety of delivering general anaesthesia to these patients.

ELIGIBILITY:
Inclusion Criteria:

* patients aged between 18 and 75 years requiring general anesthesia
* American society of Anesthesiologists (ASA) physical status classification system: I - III
* diagnosed as OSA.

Exclusion Criteria:

* Patients with chronic respiratory disease, uncontrolled hypertension, ischemic heart disease, congestive heart failure, increased intracranial pressure, gastroesophageal reflux disease,
* patients' arterial hemoglobin saturation < 98% after preoxygenation,
* patients were nasal obstruction
* patients with previous or anticipated difficult facemask ventilation or intubation,
* patients with known allergy or contraindication to propofol, remifentanil, rocuronium, or midazolam.
* patients who were unable to give informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-04-13 (Actual); Study Completion 2025-04-13 (Actual)

PRIMARY OUTCOMES:
Following the induction of general anaesthesia and muscle relaxation, the time (minutes and seconds) to peripheral oxygen saturations (SpO2) of 95%. Comparing oxygenation with THRIVE combined with nasopharyngeal or THRIVE technique. | duration from apnea to eighteen (18) minutes
  oxygenation is delivered either by THRIVE combined with nasopharyngeal or the THRIVE technique alone. General anaesthesia is induced and muscle relaxation is given. The time for the peripheral oxygen saturations (SpO2) to fall to 95% is recorded. When this occurs the trial is stopped and the patient is intubated.If 18 minutes is reached before SpO2 = 95% then the trial is stopped.

SECONDARY OUTCOMES:
Arterial partial pressure of oxygen (PaO2) | at the time apnea start, five/ten minutes after apnea and at the end of apnea
  Unit: mmHg
Arterial carbon dioxide pressure (PaCO2) | at the time apnea start, five/ten minutes after apnea and at the end of apnea
  Unit: mmHg
Concentration of arterial blood lactate | at the time apnea start, five/ten minutes after apnea and at the end of apnea
  mmol/L
Arterial blood pH | at the time apnea start, five/ten minutes after apnea and at the end of apnea
  Unitless
mininmum SPO2 | from apnea start to 1minute after intubation
  mininmum SPO2
desaturation duration(SPO2 100-99%,-98%,-95%) | from apnea start to 1minute after intubation
  desaturation duration(SPO2 100-99%,-98%,-95%)
Transcutaneous CO2 (tc CO2 increase rate | duration from apnea start to 18 minutes
  mmHg= (the tcCO2 value at the end of apnea duration minus the tcCO2 value at the beginning of the apnea duration)/apnea duration
End-tidal carbon dioxide (ETCO2) increase rate | duration from apnea start to 18 minutes
  mmHgmmHg= (the ETCO2 value at the end of apnea duration minus the ETCO2 value at the beginning of the apnea duration)/apnea duration
highest ETCO2 value ( after intubation the first PetCO2 and the highest PETCO2 among the first five) | duration from apnea start to 20 minutes
  mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Guyan Wang, Study Director — Beijing Tongren Hospital
Locations (1):
- Beijing tongren Hospital, Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Lei G, Wu L, Xi C, Yang S, Yang Q, Su S, Wang G. Apneic oxygenation with Transnasal Humidified Rapid-insufflation Ventilator Exchange (THRIVE) in obstructive sleep apnea patients: study protocol of a randomized controlled trial. BMC Anesthesiol. 2025 Apr 11;25(1):177. doi: 10.1186/s12871-025-03055-5. PMID 40217470